CLINICAL TRIAL: NCT01418950
Title: Improving Parental Knowledge: Randomized Trial of Supplementation of Prematurity Counseling With Written Information
Brief Title: Improving Parental Knowledge: Supplementation of Prematurity Counseling With Written Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00010267
Record Dates: First submitted 2010-07-26; First posted 2011-08-17 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Premature Birth
Keywords: Prematurity Counseling for pregnant women and their family
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): The control group will receive standard verbal counseling regarding outcome of premature infants
  Interventions: Other: Written information and verbal counseling
- Study Group (Experimental): Study Group will receive gestational age specific written information prior to receiving standard verbal counseling about outcome of premature infants.
  Interventions: Other: Written information and verbal counseling

INTERVENTIONS:
Other: Written information and verbal counseling — control group will only receive verbal counseling. Study group will receive written information before verbal counseling

SUMMARY:
Pregnant women who receive study counseling which includes gestational age specific written information in addition to the verbal counseling will have better knowledge of problems and outcomes of prematurity than women who receive standard counseling which consists of only verbal counseling.

ELIGIBILITY:
Inclusion Criteria:

* English speaking pregnant women who are between 23-34 weeks of gestation
* Who are 18 years and older
* Open to all ethnic groups.
* Admitted in preterm labor to Froedtert and Waukesha Hospitals labor and delivery unit.

Exclusion Criteria:

* Pregnant women who are known to have infants with congenital anomalies or other associated conditions apart from prematurity that could be a significant factor to the outcome of the baby.
* Pregnant women who have been included in this study and discharged at some point and again admitted for preterm labor will be excluded from the study.
* If a participant delivers before completing the Parent Knowledge Questionnaire, she will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maternal knowledge of problems of prematurity as measured by number of correct answers on the knowledge questionnaire will be assessed in the study and control groups. | Within 24 hours of counseling the primary outcome will be assessed
  The knowledge questionnaire consists of questions regarding gestational age specific common potential problems and complications of premature infants. We will score each questionniare and then compare number of correct answers.

SECONDARY OUTCOMES:
The change in maternal anxiety score before and after counseling as measured by the State-Trait-Anxiety-Inventory will be compared between the study and control groups | The pre-counseling anxiety score will be obtained immediately after consent is obtained for the study. The post-counseling anxiety score will be obtained within 24 hours of counseling
  State Trait anxiety Inventory has been used in many studies

CONTACTS AND LOCATIONS:
Overall Officials: Mir Basir, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Muthusamy AD, Leuthner S, Gaebler-Uhing C, Hoffmann RG, Li SH, Basir MA. Supplemental written information improves prenatal counseling: a randomized trial. Pediatrics. 2012 May;129(5):e1269-74. doi: 10.1542/peds.2011-1702. Epub 2012 Apr 9. PMID 22492766